CLINICAL TRIAL: NCT07332689
Title: A Safety Study of Quadrivalent Subunit Influenza Vaccine in a Large-Scale Population Aged 3 Years and Older
Brief Title: Safety Study of Quadrivalent Subunit Influenza Vaccine in People Aged 3 Years and Older
Status: Completed | Type: Observational
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Collaborators: Jiangsu Provincial Academy of Preventive Medicine (Unknown); Hubei Provincial Center for Disease Control and Prevention (Other); Shandong Province Centers for Disease Control and Prevention (Other); Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention (Unknown); Shanghai Municipal Center for Disease Control and Prevention (Other); Gansu Provincial Center for Disease Control and Prevention (Unknown); Guangdong Provincial Institute of Biological Products And Materia Medica (Other); Qinghai Provincial Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Other Study IDs: CDRZ20234001-2
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Influenza Vaccine
Keywords: Safety; Quadrivalent Subunit Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One dose Vaccine in aged 3 years and older
  Interventions: Biological: quadrivalent subunit influenza vaccine

INTERVENTIONS:
Biological: quadrivalent subunit influenza vaccine — one dose of quadrivalent subunit influenza vaccine

SUMMARY:
This study evaluates the safety of the quadrivalent subunit influenza vaccine following its post-marketing widespread use in individuals aged 3 years and older, aiming to assess the occurrence of very rare adverse reactions (with an incidence rate of <0.01%).

DETAILED DESCRIPTION:
This is a large-scale, multicenter, open-label, single-arm, non-controlled real-world safety observational study following influenza vaccination. It is designed to assess the occurrence of very rare adverse reactions (incidence <0.01%) following vaccination with a quadrivalent influenza subunit vaccine and to demonstrate its superior safety profile.

A total of 42,881 participants aged 3 years and above were enrolled. Each received a single 0.5 ml dose of the quadrivalent influenza subunit vaccine. Safety monitoring included immediate observation for 30 minutes post-vaccination and systematic surveillance over the subsequent 28 days. Data on adverse events (AEs) and serious adverse events (SAEs) were collected during two time intervals: from 30 minutes to 7 days (inclusive) and from 8 to 28 days (inclusive) after vaccination. Any newly identified adverse reactions during the study period were also recorded.

ELIGIBILITY:
Inclusion Criteria

1. Healthy individuals aged 3 years or above.
2. The participant (and/or their guardian/legal representative) has provided informed consent, voluntarily agreed to participate, signed the Informed Consent Form, and is able to comply with the requirements of this study protocol.

Exclusion Criteria

1. Individuals with a known allergy to any component of the vaccine, including eggs, excipients, formaldehyde, or Triton N-101.
2. Individuals suffering from an acute illness, severe chronic disease, an acute exacerbation of a chronic disease, common cold, or fever.
3. Individuals with uncontrolled epilepsy or other progressive neurological disorders, or a history of Guillain-Barré syndrome.
4. Any other condition considered by the investigator as inappropriate for participation in this study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy individuals aged 3 years or above
Sampling Method: Non-Probability Sample
Enrollment: 42881 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 30 minutes, 7 days, and 28 days after vaccination
  Occurrence of adverse events (AEs) within 30 minutes, 7 days, and 28 days after vaccination
Adverse Drug Reactions（ADR） | 30 minutes, 7 days, and 28 days after vaccination
  Incidence of known adverse drug reactions (ADRs) within 30 minutes, 7 days, and 28 days after vaccination
Serious Adverse Events (SAEs) | 28 days after vaccination
  Occurrence of serious adverse events (SAEs) within 28 days after vaccination; Incidence of new adverse reactions following vaccination

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Gansu Provincial Center for Disease Control and Prevention, Lanzhou, Gansu
  - Guangdong Provincial Institute of Biological Products and Materia Medica, Guangzhou, Guangdong
  - Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei
  - Jiangsu Provincial Academy of Preventive Medicine, Nanjing, Jiangsu
  - Qinghai Provincial Center for Disease Control and Prevention, Xining, Qinghai
  - Shandong Center for Disease Control and Prevention, Jinan, Shandong
  - Shanghai Municipal Center for Disease Control and Prevention, Shanghai, Shanghai Municipality
  - Xinjiang Uygur Autonomous Region Center for Disease Control and Prevention, Ürümqi, Xinjiang Uygur Autonomous Region